CLINICAL TRIAL: NCT00005464
Title: DISH Data Analysis Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4908; R03HL046559 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To perform extensive analyses of data from the Dietary Intervention Study of Hypertension (DISH)..

DETAILED DESCRIPTION:
BACKGROUND:

DISH was a multicenter, controlled, randomized study conducted in 1980-1983 of 496 patients, who were formerly participants in the Hypertension Detection and Follow-up Program and who had their blood pressure well controlled with medication. At DISH baseline they were randomized to continue medication or to be withdrawn from antihypertensive medication to determine if weight reduction or sodium restriction/potassium increase interventions could maintain these people under blood pressure control without drugs. Only the main findings regarding diastolic blood pressure control under the different diet regimens, were analyzed and reported during the course of DISH funding. Many questions which could be uniquely addressed by this comprehensive data base remained unexplored.

DESIGN NARRATIVE:

The investigators explored the questions dealing with demographic, clinical and physiologic predictors of relapse to the hypertensive state. They also analyzed the mortality experience of this cohort five years post DISH in relation to the DISH randomization groups and in relation to success in remaining off drugs during DISH. They did this by querying the National Death Index to determine who of the DISH participants died following the termination of DISH.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-02; Study Completion 1993-01 (Actual)

REFERENCES:
- [Background] Thaler L, Wassertheil-Smoller S, Blaufox MD, Oberman A, Langford HG. Effect of withdrawal of antihypertensive drug on depressive mood. Am J Hypertens. 1993 Dec;6(12):1055-62. doi: 10.1093/ajh/6.12.1055. PMID 8136096
- [Background] Ho GY, Blaufox MD, Wassertheil-Smoller S, Oberman A, Langford H. Plasma renin predicts success of antihypertensive drug withdrawal. Am J Hypertens. 1994 Aug;7(8):679-84. doi: 10.1093/ajh/7.8.679. PMID 7986457